CLINICAL TRIAL: NCT03927950
Title: Investigation of Genetic Predictors of the Response to SSRI Treatment
Brief Title: Investigation of Genetic Predictors of the Response to Selective Serotonin Re-uptake Inhibitors (SSRI) Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Eduard Maron, Department of Psychiatry, University of Tartu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-002649-19; 7043 (Other Grant/Funding Number: Ministry of Education, Estonia); SF0180125s08 (Other Grant/Funding Number: Ministry of Education, Estonia)
Record Dates: First submitted 2009-02-02; First posted 2019-04-25 (Actual); Results first posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Major Depression
Keywords: Treatment efficacy; Safety
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Dexetimide; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escitalopram bupropion open-label (Experimental): No comparator
  Interventions: Drug: escitalopram; Drug: bupropion

INTERVENTIONS:
Drug: escitalopram — escitalopram 10-20mg per day 12 weeks
  Other Names: Cipralex
Drug: bupropion — bupropion 150-300mg per day 6 weeks
  Other Names: Wellbutrin

SUMMARY:
The antidepressant medications are among the most commonly prescribed pharmacological agents in patients with mood and anxiety disorder. Despite recent advances in antidepressant pharmacotherapy, there is a pressing need for substantial optimization and improvment of outcome of pharmacotherapy of psychiatric disorders by providing individualized and science-based treatment guidelines. Besides it is rather difficult in clinical practice to predict, which patient will response to a certain pharmacological treatment well and which one less so. Putative predictors of response to antidepressant include demographic and clinical characteristics, personality traits, biological markers and psychophysiological features. Recently the research studies shown that divergences in antidepressant efficacy may be related to genetic variations of patients. The pharmacogenetic studies have multiplied in recent decade due to the impact that such studies may have in everyday clinical practice once reliable predictors could be identified. The pharmacogenetic research using new DNA microarray-based technology can reasonably be expected to contribute to the prediction of likelihood of treatment response and risk of development of adverse side effects in individual patients in case of antidepressant treatment. By reducing costly treatment failures and the likelihood of serious adverse events, pharmacogenetic testing may help to improve the treatment possibilities for chronic diseases, reduce the burden prescription drug costs, and lower the costs of drug development. The further detailed investigation of peripheral gene expression profiles may help to identify responsible genes that underlie the process of development of affective disorders and open novel horizons for understanding molecular mechanisms of psychopharmacological treatment.

DETAILED DESCRIPTION:
To participate in the study the subjects must be at least 18 years old and give a written informed consent after an oral and written explanation of the study aims and methods. The study sample will include the female and male patients with panic disorder or major depression diagnosis according to DSM-IV criteria. Patients will be recruited from the out- and inpatients services of the Psychiatric Clinic of the Tartu University Hospital. For the detailed assessment of clinical severity of specific disorder and treatment effects the disorder-specific rating scales: Montgomery-Asberg's Depression Rating Scale (MADRS), Clinical Global Impression scale (CGI) will be used. The adverse effects will be evaluated by letting the patients to fill the checklist of side-symptoms. In both patient groups (with panic disorder and major depression) an SSRI escitalopram (Cipralex) will be administrated for 12 weeks in flexible dose ranging between 10 - 20 mg/per day. At the end of week 12 the patients will defined as responders if the decrease in MADRS scores is at least 50% and score on the CGI improvement scale is 2 or less. The remitters will defined if the scores are less than 12 on the MADRS. Patients who do not meet these criteria will defined as non-responders and non-remitters respectively. Depressive patients, showing non-response to escitalopram monotherapy will given the combination of 20 mg of escitalopram and 150-300 mg of bupropion (Wellbutrin SR) for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Diagnosis according to DSM-IV criteria
* At severity of depression of at least moderate as indicated by a Montgomery-Asberg's Depression Rating Scale (MADRS) total score of 22 or higher
* Only secondary current comorbid anxiety disorder

Exclusion Criteria:

* Bipolar disorder
* Psychotic disorder or features
* Current eating disorders
* Mental retardation
* Any pervasive developmental disorder or cognitive disorder
* Alcohol or drug abuse-related disorders within 12 months prior to baseline
* Acute infections, neurological or any other unstable general disorders, serious suicide risk, formal behaviour therapy, or systematic psychotherapy, pregnancy or breastfeeding
* A history of hypersensitivity or non-response to escitalopram or bupropion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Maron, MD, PhD, Principal Investigator — Department of Psychiatry, University of Tartu
Locations (1):
- Department of Psychiatry, University of Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: State Agency of Medicines — http://www.ravimiamet.ee/
- See also: Department of Psychiatry — http://www.kliinikum.ee/psyhhiaatriakliinik/
- See also: University of Tartu — http://www.ut.ee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Department of Psychiatry
Groups:
- Escitalopram Bupropion Open-label: Escitalopram 10-20mg and Bupropion 150-300mg; an open-label, placebo not controlled trial in a naturalistic setting
Period: Overall Study
Arm/Group | Escitalopram Bupropion Open-label
Started | 135
Completed | 126
Not Completed | 9
Not completed — Adverse Event | 9

BASELINE CHARACTERISTICS:
Groups:
- Escitalopram: Escitalopram 10-20mg; an open-label, placebo not controlled trial in a naturalistic setting
Arm/Group | Escitalopram
Number analyzed (Participants) | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 135
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 47
Region of Enrollment [Number; unit: participants]
  Estonia | 135

OUTCOME MEASURES:

1. Secondary Outcome: Hamilton Rating Scale for Depression
Description: 17-item diagnostic questionnaire to measure the severity of depressive symptoms. The lowest possible score on the scale is 0 and the highest possible score is 52. The lowest possible score on the scale represents "the lack of any depressive symptoms" and the highest score represents the "severe depressive symptoms".
Time Frame: The outcome was measured at the week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escitalopram
Number analyzed (Participants) | 135
score on a scale | 7.2 (7.3)

2. Primary Outcome: Montgomery-Asberg's Depression Rating Scale
Description: Ten-item diagnostic questionnaire to measure the severity of depressive symptoms. The lowest possible score on the scale is 0 and the highest possible score is 60. The lowest possible score on the scale represents "the lack of any depressive symptoms" and the highest score represents the "severe depressive symptoms".
Time Frame: the results are for a single time point (12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escitalopram Bupropion Open-label
Number analyzed (Participants) | 135
score on a scale | 9.2 (10.2)

ADVERSE EVENTS:
Time Frame: During course of trial (12 weeks)
Description: 9 patients discontinued escitalopram treatment due to side effects (5 due to nausea, 4 due to sexual dysfunction)
Groups:
- Escitalopram Bupropion Open-label: Escitalopram 10-20mg Bupropion 150-300mg; an open-label, placebo not controlled trial in a naturalistic setting
Arm/Group | Escitalopram Bupropion Open-label
All-Cause Mortality (participants affected / at risk) | 0/135
Serious Adverse Events (participants affected / at risk) | 0/135
Other Adverse Events (participants affected / at risk) | 9/135
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram Bupropion Open-label (N=135)
nausea (Gastrointestinal disorders) | 5
sexual dysfunction (Reproductive system and breast disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No